CLINICAL TRIAL: NCT02054052
Title: Intrapleural Bevacizumab Injection for Treating Malignant Pleural or Pericardial Effusion in Non-small Cell Lung Cancer
Brief Title: Intrapleural Bevacizumab Injection for Malignant Effusion in Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haihong Yang, MD, Pricipal investigator (Other)
Responsible Party: Sponsor-Investigator, Haihong Yang, MD, Pricipal investigator, Deputy Chief Physician, Guangzhou Medical University
Organization: Guangzhou Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GZTO1401
Record Dates: First submitted 2014-01-27; First posted 2014-02-04 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Non-small Cell Lung Cancer; Malignant Pleural Effusion
Keywords: non-small cell lung cancer; malignant pleural effusion; bevacizumab; intrapleural injection; pericardial effusion
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pleural Effusion, Malignant; Pericardial Effusion | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Experimental): Bevacizumab 100 mg, intrapleural injection treating maliganant pleural or percardial effusion
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 100 mg, intrapleural injection treating MPE after the drainage of MPE
  Other Names: Avastin

SUMMARY:
Malignant pleural or pericardial effusion is common in lung cancer, and intrapleural drugs injection is important in the treatment. Non- cytotoxic drugs include those with a sclerosing effect that produces pleurodesis, which is easy to cause severe chest pain despite of no influence on the following chemotherapy. Tumor angiogenesis is important in producing MPE. Bevacizumab has been administrated locally in treating optic nerve sickness successfully by anti-VEGF mechanism. So we hypothesize that intrapleural bevacizumab is also effective in treating MPE.

DETAILED DESCRIPTION:
Inclusion Criteria:

1. Histological or cytological diagnosis of non-small cell lung cancer.
2. Cytological diagnosis of malignant pleural or pericardial effusion (MPE)
3. Symptomatic MPE evaluated by researchers
4. Unsuitable for or reject systemic therapy of tumor
5. Continuous TKI treatment after TKI-resistance
6. Estimated survival of more than 3 months. 7.18 years or older

Exclusion Criteria:

1. Current or recent (within 10 days prior to treatment) use the full amount of inhibition of platelet function, anticoagulants or thrombolytic therapy, which allows prophylactic anticoagulants
2. Be allergic to bevacizumab
3. Pregnant or lactating woman
4. Pleural or pericardial infection

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological diagnosis of non-small cell lung cancer.
2. Cytological diagnosis of malignant pleural or pericardial effusion (MPE)
3. Symptomatic MPE evaluated by researchers
4. Unsuitable for or reject systemic therapy of tumor
5. Estimated survival of more than 3 months. 6.18 years or older

Exclusion Criteria:

1. Current or recent (within 10 days prior to treatment) use the full amount of inhibition of platelet function, anticoagulants or thrombolytic therapy, which allows prophylactic anticoagulants
2. Be allergic to bevacizumab
3. Pregnant or lactating woman
4. Pleural or pericardial infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Lung cancer symptom | Evaluated by lung cancer symptom scale 21-30 days after the treatment

SECONDARY OUTCOMES:
response rate | Evaluate response rate 21-30 days after the treatment
Time to progression | 1 year after the treatment of MPE.
Overall survival | 1 year after the treatment of MPE
Number of Participants with Adverse Events | one months after the treatment of MPE

CONTACTS AND LOCATIONS:
Overall Officials: Haihong Yang, MD, Principal Investigator — the First Affiliated Hospital of Guangzhou MC
Locations (1):
- The First Affliliated Hospital of Guangzhou MC, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided